CLINICAL TRIAL: NCT06589947
Title: StOPping Hypertension and imprOving Children's Lives After KidnEy TranSplantation
Acronym: SOPHOCLES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Heidelberg; University of Heidelberg (Unknown); Berlin; Charité (Unknown); Bonn; Kindernieren-zentrum Bonn (Unknown); Essen; University Hospital Essen (Unknown); Frankfurt; Clementine Kinderhospital (Unknown); Hamburg; University Hospital Hamburg-Eppendorf (Unknown); Stuttgart; Olgahospital (Unknown); Hacettepe University (Other); Vienna; University Hospital Vienna (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Anette Melk, Professor of Pediatrics, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPHOCLES
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Arterial Hypertension; Kidney Transplant; Complications
Keywords: Left ventricular mass; Pediatric kidney transplantation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard BP group (Active Comparator): The treatment goal for the standard group is to achieve BP levels <90th pct.
  Interventions: Other: Standard Treatment
- Intensified BP group (Experimental): Treatment goal in the intensified group will be lowering BP ≤60th pct.
  Interventions: Other: Intensified BP control

INTERVENTIONS:
Other: Intensified BP control — Treatment goal in the intensified group will be lowering BP ≤60th pct.
  Arms: Intensified BP group
Other: Standard Treatment — Standard treatment is to achieve BP levels <90th pct.
  Arms: Standard BP group

SUMMARY:
Cardiovascular (CV) disease is a major morbidity in children after kidney transplantation (KTx), limiting life expectancy and impairing graft function. Arterial hypertension (AH) is the dominant CV risk factor, and highly abundant in this patient group. AH can cause left ventricular hypertrophy (LVH), which is predictive of CV death. LVH can be non-invasively assessed by measuring left ventricular mass index (LVMI). Analyses of observational data showed that blood pressure (BP) levels <75th percentile (pct) were associated with a significant reduction of LVMI. Guidelines give BP goals for children with chronic kidney disease (CKD). No guidelines, however, exist on the treatment of AH in pediatric KTx patients. In the proposed multicenter, randomized, parallel group trial with blinded endpoint evaluation we aim to assess n=500 pediatric patients >12 months after KTx at several KTx centers. Patients will be randomly assigned 1:1 to an intensified BP management group (BP target ≤60th pct) and a standard BP management group (BP target <90th pct). The primary endpoint is LVMI after 24 months. Secondary endpoints are estimated glomerular filtration rate (eGFR), pulse wave velocity (PWV) and intima media thickness (IMT) after 24 months. BP control will be guaranteed for both groups through BP telemonitoring, which will be transmitted in real time to the treating physician and the trial's centralized BP office. By defining the adequate BP goal, the results of the proposed study will have direct implications for the care of children after KTx. The results will define an important element of post-KTx care and help to lower CV morbidity and subsequently CV mortality of pediatric KTx patients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation >12 months ago
* Arterial hypertension

Exclusion Criteria:

* Cardiac malformation
* Treatment for a rejection episode within three months prior to inclusion

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass index (LVMI) | At 24 months after randomization
  LVMI at 24 months after randomization. Echocardiography will follow a standardized operating procedure established during the 4C study in accordance with the American Society of Echocardiography guidelines. LVMI will be calculated by dividing left-ventricular mass in grams (according to Devereux) by height in meters to the 2.16th with a correction factor of 0.09.

SECONDARY OUTCOMES:
Pulse Wave velocity (PWV) | At 24 months after randomization
  PWV at 24 months after randomization.
Estimated Glomerular Filtration Rate (eGFR) | At 24 months after randomization
  eGFR estimated by the Schwartz bedside formula at 24 months after randomization.
Intima Media Thickness (IMT) | At 24 months after randomization
  IMT at 24 months after randomization. IMT will be assessed using ultrasound with a high-resolution linear probe, by averaging five measurements from the far wall of the common carotid artery 1-2 cm proximal of the carotid bulb, following the Mannheim consensus.

OTHER OUTCOMES:
Albuminuria | At 24 months after randomization
  Albuminuria at 24 months after randomization. Albumine to creatinine ratio from spot urine will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Melk, MD PhD, Principal Investigator — Hannover Medical School

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grabitz C, Memaran N, Sugianto RI, von der Born J, Bukova M, Lehmann E, Konuhov AK, Holzwart D, Grosshennig A, Wuhl E, Schmidt BMW, Melk A. StOPping Hypertension and imprOving Children's Lives after KidnEy TranSplantation (SOPHOCLES): study protocol for a randomized controlled multicenter trial. Trials. 2025 Aug 27;26(1):315. doi: 10.1186/s13063-025-09033-z. PMID 40866927

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT06589947/Prot_SAP_000.pdf